CLINICAL TRIAL: NCT03962634
Title: Kovanaze Vs. Articaine in Achieving Pulpal Anesthesia of Maxillary Teeth: A Randomized Clinical Trial
Brief Title: Kovanaze Vs. Articaine in Achieving Pulpal Anesthesia of Maxillary Teeth - Pediatric
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug is no longer being manufactured
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20014136 - pediatric
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Results first posted 2020-11-19 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Caries,Dental; Apical Periodontitis
Keywords: Cavities
MeSH Terms: conditions — Dental Caries; Periapical Periodontitis | interventions — Tetracaine; Oxymetazoline; Carticaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Kovanaze Nasal Spray (Pediatrics) (Experimental): Children >20 kg who require pulpotomy, restorative procedures, SS crowns in one maxillary tooth
  Interventions: Drug: Kovanaze Nasal Spray
- Articaine Injections (Pediatrics) (Active Comparator): Children >20 kg who require pulpotomy, restorative procedures, or stainless steel crowns in one maxillary tooth
  Interventions: Drug: Articaine Injection

INTERVENTIONS:
Drug: Kovanaze Nasal Spray — Intra-nasal local anesthetic
  Other Names: Tetracaine HCl, Oxymetazoline HCl, NDC # 69803-100-10
  Arms: Kovanaze Nasal Spray (Pediatrics)
Drug: Articaine Injection — Local anesthetic
  Other Names: Septocaine
  Arms: Articaine Injections (Pediatrics)

SUMMARY:
The primary goal of the study is to compare the success rates of pulpal anesthesia (defined as ability to complete the intended dental procedure without the need for rescue anesthesia) between Kovanaze nasal mist and Articaine needle anesthesia.

DETAILED DESCRIPTION:
In June 2016, an intranasal delivery system of local anesthesia called Kovanaze, gained FDA approval. [9] Kovanaze is available as a 0.2 ml metered spray and is intended to achieve pulpal anesthesia of 5 maxillary teeth on either side of the face. Even though success rates between 83 and 90 % have been reported for adults and children >40kg, [10] FDA label (Section 14.2) provides data for children (>10 kg) indicating that the drug is safe for use in children as long as the dose is adjusted to bodyweight of the child. [9]

* One 0.1 mL spray for patients weighing 10 kg to less than 20 kg;
* Two 0.1 mL sprays for 20 kg to less than 40 kg; or
* Two 0.2 mL sprays for patients weighing 40 kg or more.

With the ability to avoid the traditional painful injection Kovanaze offers promise in the field of maxillary anesthesia and this study intends to:

1. Compare Kovanaze to conventional needle anesthetic children (at least 6 years of age and weighing > 20 kg)
2. Evaluate patient anxiety, tolerance and acceptability of Kovanaze in patients undergoing dental procedures

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Class I or II
* Preoperative heart rate of 55 to 100 beats per minute
* Maximum blood pressure reading of 166/100 mmHg
* Treatment for a pathology in the maxillary anterior tooth or premolar that requires administering local anesthesia

Additional Pediatric Inclusion Criteria:

* Children >20 kg who require pulpotomy, restorative procedures, or stainless steel crowns in one maxillary tooth

Additional Endodontic Inclusion Criteria:

* Adults (>18 years) who require non-surgical root canal treatment in maxillary anterior teeth

Additional General Practice Inclusion Criteria:

* Adults who require restorations in the maxillary teeth that would need local anesthesia

Exclusion Criteria:

* Inadequately controlled thyroid disease
* Five or more nosebleeds in the past month
* Known allergy to any study drug or para-aminobenzoic acid
* History of methemoglobinemia
* Taking monoamine oxidase inhibitors, tricyclic antidepressants (i.e. amitriptyline), or non-selective beta adrenergic antagonists (i.e. propranolol);
* Taking oxymetazoline-containing products (i.e., Afrin) in the last 24 hours.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-28 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Parthasarathy Madurantakam, DDS, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because of the low number of enrollees with only 1 in the treatment group, results are not reported to protect the confidentiality of the participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics) | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Because of the low number of enrollees with only 1 in the treatment group, results are not reported to protect the confidentiality of the participants
Sex: Female, Male [Count of Participants; unit: Participants] — Because of the low number of enrollees with only 1 in the treatment group, results are not reported to protect the confidentiality of the participants Population: Because of the low number of enrollees with only 1 in the treatment group, results are not reported to protect the confidentiality of the participants
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Pupal Anesthesia
Description: % dental procedures completed without the need for rescue anesthesia
Time Frame: immediately after dental procedure, an average of 3 hours
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Spread of Anesthesia
Description: Number of teeth anesthetized in maxillary arch
Time Frame: immediately after dental procedure, an average of 3 hours
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Anxiety Level
Description: STAI-Y6 - 6 item youth questionnaire assessing anxiety on a 4 point scale ranging from 1 (Not at all) to 4 (very much). Scores range from 6 to 24.
Time Frame: from baseline to immediately after dental procedure
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Anxiety
Description: Venham Behavior rating scale - single item 6 point scale used by provider to rate child's behavior during treatment. Item ranges from 0 (no protest) to 5 (high protest, no cooperation from child)
Time Frame: immediately after dental procedure, an average of 3 hours
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Blood Pressure
Time Frame: from baseline to immediately after dental procedure
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Heart Rate
Time Frame: from baseline to immediately after dental procedure
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Pain
Description: Emoji scale ranging from 1 (very negative face) to 7 (very positive face)
Time Frame: from baseline to immediately after dental procedure
Population: as for baseline characteristics
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 3 hours, the length of the dental procedure
Arm/Group | Kovanaze Nasal Spray (Pediatrics) | Articaine Injections (Pediatrics)
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/34/NCT03962634/Prot_SAP_002.pdf